CLINICAL TRIAL: NCT03180788
Title: The Impact of Traction Assisted ESD on Procedural Time, En Bloc Resection, Curative Resection and Complication Incidence
Brief Title: The Impact of Traction Assisted ESD on Procedural Time and Outcome
Acronym: ESD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was never started
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLIPTHREAD
Record Dates: First submitted 2017-05-30; First posted 2017-06-08 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Colorectal Polyp
Keywords: ESD; Traction assisted ESD; Polypectomy; Clip and thread ESD

STUDY DESIGN:
Intervention Model Description: Prospective randomiced Clinical trial
Who Masked: Investigator
Masking Description: Randomisation to either traction assisted ESD or traditional ESD
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional ESD (Active Comparator): The patients in this Group will undergo traditional ESD.
  Interventions: Procedure: Traditional ESD
- Traction assisted ESD (Experimental): The patients in this Group will undergo traction assisted ESD
  Interventions: Procedure: Traction assisted ESD

INTERVENTIONS:
Procedure: Traction assisted ESD — A clip attached to a thread is mounted on the lesion. Traction is achieved by pulling the thread during ESD
  Arms: Traction assisted ESD
Procedure: Traditional ESD — Endoscopic submucosa dissection
  Arms: Traditional ESD

SUMMARY:
The aim of this study is to evaluate the role of traction assisted ESD in comparison to traditional ESD on procedural time and outcome in patients with large, non pedunculated colorectal polyps.

DETAILED DESCRIPTION:
Endoscopic polypectomy, has been proven to reduce Colorectal cancer incidence and mortality. Smaller lesions and pedunculated lesions can be removed by conventional polypectomy, Endoscopic mucosa resection (EMR). However, large sessile and flat lesions are difficult to remove En bloc with EMR, resulting in a high level of tumor recurrence. Endoscopic submucosal dissection (ESD) was developed during the 1990s in Japan to achieve En bloc resection of large neoplasms in the stomach but has in recent years also been extended into management of large (>2 cm) and technically challenging colorectal polyps. Large series on the efficacy of ESD in removing benign lesions show high En bloc resection rates resulting in low numbers of recurrences. Traction assisted ESD was developed in Japan to further improve the technique and reduce procedural time, the literature on the efficacy of traction assisted ESD is however scarce and limited to Japanese studies.

The aim in this study is to investigate the impact of this novel technique in comparison to traditional ESD on procedural time, En bloc resection rate, R0 resection rate and complication incidence.

ELIGIBILITY:
Inclusion Criteria:

* > 2cm, flat or sessile colorectal polyp

Exclusion Criteria:

* Recurrencies.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-08 (Estimated); Primary Completion 2018-12-20 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Procedural time | 280 min, procedural time
  Time consumption to complete the resection is measured.

SECONDARY OUTCOMES:
En bloc resection | 280 min, procedural time
  En bloc resection rates will be recorded
R0 resection | 4-8 weeks, when pathological examination is completed
  R0 resection rate, stated in the pathology report will be recorded
Complication incidence | 2 weeks, when the timeframe for delayed complications is over.
  All complications both immediate and delayed will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Skane University Hospitals, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saito Y, Uraoka T, Yamaguchi Y, Hotta K, Sakamoto N, Ikematsu H, Fukuzawa M, Kobayashi N, Nasu J, Michida T, Yoshida S, Ikehara H, Otake Y, Nakajima T, Matsuda T, Saito D. A prospective, multicenter study of 1111 colorectal endoscopic submucosal dissections (with video). Gastrointest Endosc. 2010 Dec;72(6):1217-25. doi: 10.1016/j.gie.2010.08.004. Epub 2010 Oct 27. PMID 21030017
- [Result] Ritsuno H, Sakamoto N, Osada T, Goto SP, Murakami T, Ueyama H, Mori H, Matsumoto K, Beppu K, Shibuya T, Nagahara A, Ogihara T, Watanabe S. Prospective clinical trial of traction device-assisted endoscopic submucosal dissection of large superficial colorectal tumors using the S-O clip. Surg Endosc. 2014 Nov;28(11):3143-9. doi: 10.1007/s00464-014-3572-0. Epub 2014 May 31. PMID 24879138